CLINICAL TRIAL: NCT00930332
Title: A Phase I Study to Determine the Dose of Methadone as a First Line Agent in the Treatment of Chronic Neuropathic Cancer Pain
Brief Title: Methadone Hydrochloride as First-Line Therapy in Treating Patients With Chronic Neuropathic Cancer Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SC22; CAN-NCIC-SC22 (Registry Identifier: PDQ); CDR0000641372 (Other: PDQ)
Record Dates: First submitted 2009-06-27; First posted 2009-06-30 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2020-04

CONDITIONS: Nausea and Vomiting; Pain; Sleep Disorders; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: sleep disorders; nausea and vomiting; unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Nausea; Vomiting; Pain; Sleep Wake Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Methadone (Active Comparator): Level 1: 1 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA** per day)
  Level 2: 2 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 3: 3 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Interventions: Drug: methadone hydrochloride; Other: questionnaire administration; Procedure: management of therapy complications
- Arm B: Methadone (Active Comparator): Level 1: 2 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 2: 3 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 3: 4 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Interventions: Drug: methadone hydrochloride; Other: questionnaire administration; Procedure: management of therapy complications

INTERVENTIONS:
Drug: methadone hydrochloride — Level 1: 1 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA** per day)
  Level 2: 2 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 3: 3mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  OR
  Level 1: 2 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 2: 3 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
  Level 3: 4 mg q8h, breakthrough 1 mg q2h* (maximum 6 BTA per day)
Other: questionnaire administration — within 48 hours of registration
Procedure: management of therapy complications — if required

SUMMARY:
RATIONALE: Methadone hydrochloride may reduce chronic neuropathic pain in patients with cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of methadone hydrochloride as first-line therapy in treating patients with chronic neuropathic cancer pain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the optimum starting dose (defined as the dose that does not require modification within the first 4 days of treatment for lack of efficacy or the occurrence of adverse events) of methadone hydrochloride as a first-line opioid treatment in patients with chronic neuropathic cancer pain.

Secondary

* To assess the number and timing of breakthrough analgesic usage.
* To assess the number of episodes of breakthrough pain.
* To assess the total daily dose of methadone hydrochloride.
* To assess the average pain score.
* To determine the safety and adverse event profile of methadone hydrochloride as a first-line opioid in the treatment of chronic neuropathic cancer pain.
* To assess the frequency and severity of sleep disturbance associated with the use of methadone hydrochloride.
* To determine the feasibility of recruiting patients with chronic neuropathic cancer pain in a reasonable time frame for a future phase III study of methadone hydrochloride vs morphine.

OUTLINE: This is a multicenter study. Patients are assigned to a group according to their average daily dosage of morphine-equivalent for the 3 full days prior to study entry (≤ 45 mg/day OR > 45 but ≤ 75 mg/day).

Patients receive oral methadone hydrochloride at various doses every 8 hours. Patients also may receive breakthrough oral methadone hydrochloride every 2 hours, as needed, for up to 6 breakthrough analgesics per day. Treatment continues for up to 35 days. Treatment stops if the patient has well-controlled pain or experiences intolerable side effects.

Patients complete the Short-Form McGill Pain Questionnaire at baseline. Patients rate their pain according to questions from the Brief Pain Inventory on a scale of 0 (no pain) to 10 (worst pain imaginable) to best describe pain at its worst in the last 24 hours, pain at its least in the last 24 hours, pain on average, and pain right now; record the number and timing of breakthrough analgesic usage, the number of episodes of breakthrough pain, and the total daily dose of methadone hydrochloride; and complete nausea and sleep assessments once daily on days 1-14.

After completion of study treatment, patients are followed at 4, 6-7, and 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients diagnosed with cancer and experiencing chronic neuropathic pain syndrome

  * Pain syndrome diagnosed by the investigator
  * Pain syndrome related to the effects of cancer or its treatment (i.e., chemotherapy, radiotherapy, and surgery)
  * Meets 1 of the following criteria:

    * Need to be started on strong opioids
    * Require an increase in opioid dose and are currently taking ≤ 75 mg of total daily dose of oral morphine equivalent
* Experiencing pain for ≥ 4 weeks with an average pain score of ≥ 4 or a worst pain score of ≥ 5 (using the 0-10 Brief Pain Inventory Scale) during the past 24 hours
* Requires strong opioids to control pain and is using an oral morphine-equivalent dose of 0-75 mg per day, on average, including breakthrough analgesia, within the past 3 full calendar days
* Mixed pain syndrome allowed provided the neuropathic component is the predominant pain
* Meets 1 of the following criteria:

  * Receiving concurrent chemotherapy but the chronic neuropathic pain is not related to this treatment and is not expected to improve or worsen because of this therapy
  * Received prior chemotherapy but discontinued treatment, has not received chemotherapy within the past 7 days, and no further chemotherapy is planned
  * No prior chemotherapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 40-100%
* ALT and AST ≤ 3 times upper limit of normal (ULN)
* Creatinine ≤ 2 times ULN
* No other known laboratory abnormality that, in the investigator's opinion, would contraindicate study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Mini-Mental State Examination score ≥ 25/30
* Able to speak, read, and write in either English or French
* Willing to complete study diary and questionnaires
* Available for study treatment and follow up (i.e., within reasonable geographical limits of the participating center)
* Able to swallow and tolerate oral medications
* Patients with prior exposure to methadone hydrochloride must be able to tolerate it
* No intractable nausea and vomiting
* No presence or history of unstable disease or condition that would, in the investigator's opinion, preclude patient participation in study treatment, such as:

  * Head injury
  * Increased intracranial pressure
  * Uncontrolled seizures
  * Uncontrolled asthma
  * Decompensated chronic obstructive pulmonary disease
  * Untreated prostate hypertrophy
  * Acute abdominal conditions
  * Untreated hyperthyroidism and Addison disease
  * Increased cerebrospinal fluid pressure
  * Urethral stricture
  * Severe cardiac arrhythmias (especially prolonged QT interval)
  * Symptomatic hypotension
  * Toxic psychosis
  * Cor pulmonale
  * Sleep apnea
  * Severe obesity
  * Kyphoscoliosis
  * Myxedema
  * Central nervous system depression
  * Coma
* No history of significant alcohol, analgesic, or narcotic substance abuse within the past 6 months
* Able physically and mentally to answer questions and comply with study treatment
* No patient who lives alone and cannot access at least 1 caregiver who can monitor on a daily basis at home

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior radiopharmaceutical treatment or radiotherapy
* Concurrent co-analgesics and medications that can affect methadone hydrochloride metabolism allowed provided patients have been on a stable dose for the past 3-5 days and ≥ 5 half lives have passed since any change in dose
* Not scheduled to start chemotherapy during the study treatment
* Not planning on starting or discontinuing medication associated with modified methadone hydrochloride clearance during study treatment
* No concurrent therapeutic procedure that is likely to influence pain intensity during the study period
* No concurrent other opioid medications
* No other concurrent methadone hydrochloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06-17 (Actual); Primary Completion 2012-01-06 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Optimum starting dose | 28 days

SECONDARY OUTCOMES:
Pain control as assessed by the number and timing of breakthrough analgesics, the number of episodes of breakthrough pain, the total daily dose of methadone, and the average pain scores | 28 days
Adverse events (including respiratory depression) according to NCI CTCAE v3.0 criteria | 28 days
Frequency and severity of sleep disturbance from pain | 28 days
Feasibility of recruiting patients | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gagnon, MD, MSC, Study Chair — McGill Cancer Centre at McGill University; Ray Viola, Study Chair — Queen's University
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No